CLINICAL TRIAL: NCT03154671
Title: Clinical and Cost-effectiveness of a Comprehensive Geriatric Assessment and Management for Canadian Elders With Cancer: the 5C Study
Brief Title: Comprehensive Geriatric Assessment and Management for Canadian Elders With Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toronto (Other)
Collaborators: University Health Network, Toronto (Other); The Ottawa Hospital (Other); Sir Mortimer B. Davis - Jewish General Hospital (Other); R.S. McLaughlin Durham Cancer Centre, Lakeridge Health (Unknown); Sunnybrook Health Sciences Centre (Other); Fraser Health (Other); Mount Sinai Hospital, Canada (Other)
Responsible Party: Principal Investigator, Martine Puts, Assistant Professor, University of Toronto
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 705046
Record Dates: First submitted 2017-05-10; First posted 2017-05-16 (Actual); Last update posted 2022-05-20 (Actual); Status verified 2022-05

CONDITIONS: Cancer
Keywords: older adult;; comprehensive geriatric assessment; chemotherapy; integrated care; randomized controlled trial
MeSH Terms: conditions — Neoplasms | interventions — Geriatric Assessment; Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The outcome assessor and statistician will be blinded to group allocation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): At study enrollment participants allocated to the intervention arm will complete a comprehensive geriatric assessment with the study intervention team (nurse and physician). Based on these findings a care plan tailored to the needs of the older adult with cancer will be developed and implemented. The study intervention nurse will call the participant at least monthly to follow up and evaluate the care (e.g. whether adjustments are required) and more if needed. All participants will receive a monthly healthy aging newsletter.
  Interventions: Other: Geriatric assessment and management
- Control group (No Intervention): The participant will receive usual care from their treating oncology team. All participants will receive a monthly healthy aging newsletter.

INTERVENTIONS:
Other: Geriatric assessment and management — Each participant will receive a comprehensive geriatric assessment at baseline. Based on the issues identified, a tailored care plan will be developed with the participant to address the issues identified.
  Arms: Intervention group

SUMMARY:
A multicentre two-group parallel single-blind (outcome assessor) randomized controlled trial (RCT). A cost effectiveness study alongside a clinical trial using a payer and societal perspective to study the cost-effectiveness of geriatric assessment and management compared to usual care will be conducted.

Participants allocated to the control group will receive usual oncology care. Participants allocated to the intervention group will receive a comprehensive geriatric assessment and management in addition to their usual oncology care. The intervention will take 6 months to be completed. Total study follow-up will be 12 months for each participant.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 70+ with any solid tumor (excluding pancreatic) or lymphoma/myeloma referred for first/second line adjuvant/curative or palliative chemotherapy (cannot have received more than 1 cycle),
* Able to speak English/French,
* Have a physician-estimated life expectancy >6 months,
* Have an ECOG Performance Score 0-2 (indicating participants are ambulatory and able to complete all self-care activities),
* Able to give informed consent.

Exclusion Criteria:

* Receiving palliative care services upon recruitment
* Already participating in another psychosocial/educational intervention study (new treatment study is allowed if the participants would like to participate in 2 studies)

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 351 (Actual)
Dates: Start 2018-04-10 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-04-01 (Actual)

PRIMARY OUTCOMES:
Quality of Life questionnaire (QLQ) C30 Questionnaire Global quality of Life scale | 6 months
  Quality of Life questionnaire (QLQ) C30 Questionnaire Global quality of Life scale
Quality of Life questionnaire (QLQ) C30 Questionnaire Global quality of Life scale | 12 months
  Quality of Life questionnaire (QLQ) C30 Questionnaire Global quality of Life scale

SECONDARY OUTCOMES:
Cost-effectiveness | 12 months
  Cost-effectiveness will be determined alongside the clinical trial following standard guidelines. 2 methods to collect data needed for the cost-effectiveness analyses: 1) EQ-5D-5L and 2) patient health care use diaries
Functional status | 6 months
  Instrumental Activities of Daily Living (OARS IADL questionnaire)
Functional status | 12 months
  Instrumental Activities of Daily Living (OARS IADL questionnaire)
The number of geriatric issues successfully addressed for participants in intervention group | 6 months
  The number of referrals/recommendations made to the participant and the number implemented by the participant
Treatment toxicity | 6 months
  Grade 3-5 chemotherapy treatment toxicity using the Common Terminology Criteria for Adverse Events v4.0 (CTCAE)[12] and treatment completion rate (number of cycles received) will be abstracted from the medical chart
Unplanned health care use | 6 months
  Unplanned hospitalization and emergency department visits abstracted from patient diary and medical chart
Satisfaction with care provided | 6 months
  Older adult and medical oncologists will be asked to rate their satisfaction with the intervention
Satisfaction with intervention | 12 months
  Older adult and medical oncologists will be asked to rate their satisfaction with the intervention
Cancer treatment plan modification | 3 months
  Whether the medical oncologist changed the treatment plan after receiving the geriatric assessment results
Overall survival | 12 months
  Overall survival will be abstracted from the medical chart
Intervention fidelity by treatment centre | 12 months
  A detailed process evaluation looking at the implementation of the intervention by centre will be conducted

CONTACTS AND LOCATIONS:
Overall Officials: Martine Puts, RN PhD, Principal Investigator — University of Toronto
Locations (2):
- Canada (2):
  - Lakeridge Health, Oshawa, Ontario
  - Princess Margaret Cancer Centre, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Habib MH, Alibhai SMH, Puts M. How representative are participants in geriatric oncology clinical trials? The case of the 5C RCT in geriatric oncology: A cross-sectional comparison to a geriatric oncology clinic. J Geriatr Oncol. 2024 Mar;15(2):101703. doi: 10.1016/j.jgo.2024.101703. Epub 2024 Jan 15. PMID 38228054
- [Derived] Puts M, Alqurini N, Strohschein F, Koneru R, Szumacher E, Mariano C, Monette J, Hsu T, Brennenstuhl S, McLean B, Wills A, Berger A, Amir E, Romanovsky L, Li A, Mehta R, Krzyzanowska M, Elser C, Jang R, Prica A, Wan-Chow-Wah D, Pitters E, Emmenegger U, Menjak IB, Bergman S, Lemonde M, Breunis H, Beland F, Alibhai SMH. Impact of Geriatric Assessment and Management on Quality of Life, Unplanned Hospitalizations, Toxicity, and Survival for Older Adults With Cancer: The Randomized 5C Trial. J Clin Oncol. 2023 Feb 1;41(4):847-858. doi: 10.1200/JCO.22.01007. Epub 2022 Dec 6. PMID 36473126
- [Derived] Puts MTE, Hsu T, Mariano C, Monette J, Brennenstuhl S, Pitters E, Ray J, Wan-Chow-Wah D, Kozlowski N, Krzyzanowska M, Amir E, Elser C, Jang R, Prica A, Krahn M, Beland F, Bergman S, Koneru R, Lemonde M, Szumacher E, Zidulka J, Fung S, Li A, Emmenegger U, Mehta R, Flemming K, Breunis H, Alibhai SMH. Clinical and Cost-effectiveness of a Comprehensive geriatric assessment and management for Canadian elders with Cancer-the 5C study: a study protocol for a randomised controlled phase III trial. BMJ Open. 2019 May 10;9(5):e024485. doi: 10.1136/bmjopen-2018-024485. PMID 31079079